CLINICAL TRIAL: NCT02042677
Title: User Assessment of a One-Piece Skin Barrier
Brief Title: Assessment of a Skin Barrier
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment of participants
Sponsor: Hollister Incorporated (Industry)
Collaborators: St George's Healthcare NHS Trust (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5566-O
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Ileostomy
Keywords: ileostomy; 1-piece; assessment; Nova; NovaLife; Dansac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This evaluation is being conducted to determine user perception of a new flat one-piece skin barrier compared to their normal barrier.

DETAILED DESCRIPTION:
Design:

This is a multi-site, unblinded, historically controlled assessment of a one-piece flat skin barrier. Study barriers are CE-marked. Approximately 30 subjects are enrolled in the UK.

ELIGIBILITY:
Inclusion Criteria:

1. is at least 18 years of age.
2. has an ileostomy.
3. is at least six weeks postoperative.
4. lives and cares for their stoma independently in the community.
5. currently uses a Dansac Nova or NovaLife 1-piece flat skin barrier.
6. currently uses a drainable pouch.
7. is able to wear a 1-piece flat cut-to-fit 10-55 mm.
8. Has a peristomal skin irritation score of 2 or less.
9. is willing to follow the protocol as demonstrated by signing the informed consent and who in the opinion of the investigator is qualified to participate.

Exclusion Criteria:

1. has a fistula on or near the stoma.
2. has been involved in a study involving stoma care with in the last 30 days.
3. is pregnant or lactating, as determined by interview only.
4. is undergoing chemotherapy, radiation or steroid therapy.
5. has an existing medical condition that would compromise their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current users of either Dansac flat Nova or NovaLife skin barriers with drainable pouches who have an ileostomy.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
barrier adhesion | 10 days
  Questionnaire will be provided to subject to assess barrier adhesion.
barrier tack | 10 days
  Questionnaire will be provided to subject to assess barrier tack.
comfort | 10 days
  Questionnaire will be provided to subject to assess comfort.
leakage | 10 days
  Questionnaire will be provided to subject to assess leakage.
ease of barrier removal | 10 days
  Questionnaire will be provided to subject to assess ease of barrier removal.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Dennis, Principal Investigator — St. George's Hospital; Sarah Varma, Stoma Nurse, Principal Investigator — St. Mark's Hospital
Locations (2):
- United Kingdom (2):
  - St. Mark's Hospital, Harrow
  - St. George's Hospital, London